CLINICAL TRIAL: NCT02009111
Title: Dyadic, Skills-Based Primary Prevention for Partner Violence in Perinatal Parents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 7U49CE001246-06 (NIH)
Record Dates: First submitted 2013-11-15; First posted 2013-12-11 (Estimated); Last update posted 2022-11-02 (Actual); Status verified 2013-12

CONDITIONS: Intimate Partner Violence
Keywords: Transition to parenthood; Relationship intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Couple CARE for Parents (Experimental): Couple CARE for Parents is a couple-focused intervention that addresses interpersonal processes within relationships and promotes healthy relationship and parenting skills among couples with a newborn. Couple CARE for Parents uses a highly disseminable model (i.e., home-visitation and video- and telephone-assisted skills training) developed in Australia.
  Interventions: Behavioral: Couple CARE for Parents
- Wait-list control (Other): The control group will be wait-listed until after the 24-month assessment, at which point they are eligible to receive Couple CARE for Parents (tailored for their children's ages).
  Interventions: Behavioral: Couple CARE for Parents

INTERVENTIONS:
Behavioral: Couple CARE for Parents — Couple CARE for Parents is a skill-based relationship enhancement program based on a self-regulatory model. It consists of seven sessions and two follow-up booster sessions that occur over the baby's first eight months of life. The first home visit is scheduled 7 - 14 days following recruitment. The next two sessions are scheduled in two week intervals. Sessions 4 through 7 are scheduled in three week intervals. Home visits are expected to last 1.5 to 2 hrs. Out-of-session viewing of the video and completing the exercises typically requires 45 min to 1 hr. The typical phone consultation lasts 15- to 30- min per person. Thus, the program lasts a minimum of 8 to 12 hours. The program will also include two booster sessions (beyond the 8 - 12 hrs).

SUMMARY:
Couple CARE for Parents is a couple-focused intervention that addresses interpersonal processes within relationships and promotes relationship and parenting skills among couples with a newborn. Couple CARE for Parents uses an approach developed in Australia that was designed to be fairly easy and cost-effective to disseminate widely (i.e., home-visitation and video- and telephone-assisted skills training). It has demonstrated efficacy for significantly enhancing couples' relationship satisfaction in three Australian randomized trials.

Arresting the normal decline of satisfaction of new parents to near-clinical levels is noteworthy because relationship dissatisfaction is one of the strongest predictors of partner physical assault. Managing relationship conflict is critical to the health and well-being of both parents and their children. Given the high prevalence of partner physical and emotional aggression (a precursor to the more serious form labeled "intimate partner violence" [IPV]) in new parents) among perinatal parents, the need for efficacious prevention services is acute.

This randomized, controlled trial will test if couples with a newborn who receive Couple CARE for Parents report significantly less IPV than control couples who do not receive the program. This is a prevention trial. No couple will report ever having experienced IPV. All couples will have three empirically documented risk factors for the development of IPV: youth (each couple will have at least one partner under 30 years of age), parenting a newborn, and psychological aggression in the past year.

The project has the following aims: (1) Determine the outcomes of Couple CARE for Parents. The investigators hypothesize that, among other positive outcomes, couples who receive Couple CARE for Parents, compared with those who do not, will report at follow-up (a) less IPV; and (b) less partner physical and emotional aggression. (2) Identify factors that may contribute to reduction in IPV and in physical and emotional aggression (e.g., communication skills, conflict behaviors, parenting expectations, , quality of adult attachment, partner attributions, child abuse potential, family income, marital status, parenting stress, infant difficultness).

ELIGIBILITY:
Inclusion Criteria:

* Couples are the unit of inclusion. Thus, individuals must be in a relationship. The following criteria are at the couple level.
* must be living together
* must have at least one member aged 30 years or younger
* must have a baby less than 3 months of age at the time of enrollment
* must have at least one member who, based on self- or partner-report, has been verbally or psychologically aggressive in the previous six months
* have two partners able to complete assessments in English
* have never engaged in intimate partner violence, by both partners' reports

Exclusion Criteria:

* Any of the above not met.
* One member less than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 706 (Actual)
Dates: Start 2008-03; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Conflict Tactics Scale Change from Assessment 1 to Assessment 2 | Assessment 1 (0-3 months); Assessment 2 (8 months)
  The CTS2 is a 78-item inventory that assesses the frequency (on 0 - 6 scales labeled from "never" to "more than 20 times") of perpetration of and victimization by partner conflict behaviors in the past 6 months.
Conflict Tactics Scale Change from Assessment 1 to Assessment 3 | Assessment 1 (0-3 months); Assessment 3 (15 months)
  The CTS2 is a 78-item inventory that assesses the frequency (on 0 - 6 scales labeled from "never" to "more than 20 times") of perpetration of and victimization by partner conflict behaviors in the past 6 months.
Conflict Tactics Scale Change from Assessment 1 to Assessment 4 | Assessment 1 (0-3 months); Assessment 4 (24 months)
  The CTS2 is a 78-item inventory that assesses the frequency (on 0 - 6 scales labeled from "never" to "more than 20 times") of perpetration of and victimization by partner conflict behaviors in the past 12 months.

SECONDARY OUTCOMES:
Child Abuse Potential Inventory Change from Assessment 1 to Assessment 2 | Assessment 1 (0-3 months); Assessment 2 (8 months)
  This 70-item self-report measure contains 70 of the original 77 abuse items.
Infant Difficultness Questionnaire Change from Assessment 1 to Assessment 2 | Assessment 1 (0-3 months), Assessment 2 (8 months)
  This is a 24-item parent-report measure of perceived difficult temperament.
Couples Satisfaction Index Change from Assessment 1 to Assessment 2 | Assessment 1 (0-3 months), Assessment 2 (8 months)
  This is a measure of relationship satisfaction.
Child Abuse Potential Inventory Change from Assessment 1 to Assessment 3 | Assessment 1 (0-3 months); Assessment 3 (15 months)
  This 70-item self-report measure contains 70 of the original 77 abuse items.
Child Abuse Potential Inventory Change from Assessment 1 to Assessment 4 | Assessment 1 (0-3 months); Assessment 4 (24 months)
  This 70-item self-report measure contains 70 of the original 77 abuse items.
Infant Difficultness Questionnaire Change from Assessment 1 to Assessment 3 | Assessment 1 (0-3 months); Assessment 3 (15 months)
  This is a 24-item parent-report measure of perceived difficult temperament.
Infant Difficultness Questionnaire Change from Assessment 1 to Assessment 4 | Assessment 1 (0-3 months); Assessment 4 (24 months)
  This is a 24-item parent-report measure of perceived difficult temperament.
Couples Satisfaction Index Change from Assessment 1 to Assessment 3 | Assessment 1 (0-3 months); Assessment 3 (15 months)
  This is a measure of relationship satisfaction.
Couples Satisfaction Index Change from Assessment 1 to Assessment 4 | Assessment 1 (0-3 months); Assessment 4 (24 months)
  This is a measure of relationship satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- New York University, New York, New York, United States

REFERENCES:
- [Background] Petch JF, Halford WK, Creedy DK, Gamble J. A randomized controlled trial of a couple relationship and coparenting program (Couple CARE for Parents) for high- and low-risk new parents. J Consult Clin Psychol. 2012 Aug;80(4):662-73. doi: 10.1037/a0028781. Epub 2012 Jun 25. PMID 22730950
- [Background] Halford WK, Sanders MR, Behrens BC. Can skills training prevent relationship problems in at-risk couples? Four-year effects of a behavioral relationship education program. J Fam Psychol. 2001 Dec;15(4):750-68. doi: 10.1037//0893-3200.15.4.750. PMID 11770479
- [Background] Halford WK; Moore EM; Wilson KL; Dyer C; Farrugia C. Benefits of a flexible delivery relationship education: An evaluation of the Couple CARE program. Fam Relat 2004 June;53:469-476